CLINICAL TRIAL: NCT01502566
Title: A Cluster-randomized Trial of the Effectiveness of an Educational Intervention in Preventing Early Childhood Caries
Brief Title: Educational Intervention in Preventing Early Childhood Caries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, PhD, Associate Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UFPEL-PPGO0011
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Dental Caries
Keywords: educational intervention; dentals caries; population; new populational caries prevention strategies.
MeSH Terms: conditions — Dental Caries | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention (Experimental): Children/mothers allocated to this arm will receive an pamphlet with key information on dental caries prevention, together with oral instructions about how to avoid dental caries. This intervention will be applied at the Brazilian National Vaccination Day
  Interventions: Behavioral: Education Intervention
- Control group (No Intervention): This group will receive no intervention

INTERVENTIONS:
Behavioral: Education Intervention — Children/mothers allocated to this arm will receive an pamphlet with key information on dental caries prevention, together with oral instructions about how to avoid dental caries.
  Arms: Educational Intervention

SUMMARY:
Objective:

The aim of this study is to assess the effectiveness of an oral health educative intervention in preventing early childhood caries (ECC).

Methods:

The trial targets 0- to 12-month-old children and their mothers in Pelotas, Brazil. Twenty-four public health centres (clusters) were randomly selected and assigned to intervention or control group (12 clusters per intervention group). In each center, up to 30 children/mothers were selected and invited to participate in the trial. Each mother was interviewed in order to collect socio-economic and demographic variables. The intervention group received by means of a pamphlet the oral health instructions, which were emphasized with verbal instructions. Dental examination will be carried out after 1 year for all teeth surfaces to determine caries status.

ELIGIBILITY:
Inclusion Criteria:

* Children with 0 to 12 months

Exclusion Criteria:

* Children with teeth in mouth at the time of enrollment
* Children not living in Pelotas
* No sufficient information provided by the mother at the time of enrollment
* Systemic diseases

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Caries status (dmfs) | after 12 months
  Number of carious lesions, including intial lesions (white spot), per surface teeth. Also missed and filled surfaces due to caries will be included.

SECONDARY OUTCOMES:
dental plaque index | after 12 months
  The oral health status will be recorded by visible dental plaque index.

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano S Cenci, PhD, Principal Investigator — Federal University of Pelotas; Marina S Azevedo, MSc, Principal Investigator — Federal University of Pelotas; Ana R Romano, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas - School of Dentistry, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed?term=mohebbi%202009%20caries